CLINICAL TRIAL: NCT06750276
Title: A Phase 2a, Randomised, Single-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics and Explore the Pharmacodynamic Effects of AZD2389 in Participants With Liver Fibrosis and Compensated Cirrhosis
Brief Title: A Study to Evaluate the Safety, Tolerability, PK, and PD Effects of AZD2389 in Participants With Liver Fibrosis and Compensated Cirrhosis.
Acronym: BORANA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D7930C00002
Record Dates: First submitted 2024-12-06; First posted 2024-12-27 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Liver Fibrosis; Hepatic Cirrhosis
Keywords: Liver Fibrosis; Hepatic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: The total duration of study participation for each participant in Cohorts A and B will be approximately 63 days (9 weeks) and will include an up to 28-day screening period, a 28-day treatment period, and a follow-up visit seven days following completion of treatment.
  Assessments will be conducted as described in the SoA.
Who Masked: Participant, Investigator
Masking Description: This is a single-blind, randomized, placebo-controlled study with up to 2 study intervention cohorts that are participant and investigator-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Other): Participants with presumed MASH/NASH with fibrosis will be screened such that approximately 18 participants will be randomised. Twelve participants will be randomised to receive AZD2389 and 6 participants will receive placebo.
  Interventions: Drug: AZD2389
- Cohort B (Other): Participants with SLD with advanced fibrosis including compensated cirrhosis will be screened such that approximately 18 participants will be randomised. Twelve participants will be randomised to receive AZD2389 and 6 participants will receive placebo.
  Interventions: Drug: AZD2389

INTERVENTIONS:
Drug: AZD2389 — Doses of AZD2389 or placebo will be administered orally.

SUMMARY:
The purpose of this study is to measure the safety, tolerability, and the way the body absorbs, distributes, and metabolises AZD2389 as compared to placebo in participants with liver fibrosis and compensated cirrhosis. The study will also examine how the drug acts on the body

DETAILED DESCRIPTION:
Study details include:

The study duration will be up to 63 days (9 weeks).

* 1 or 2 screening visits (up to 28 days before treatment)
* 28 days of treatment including 5 clinic visits
* Week 1: 24-hour in-clinic stay (Day 1)
* Week 2: Outpatient clinic visit (Day 7)
* Week 3: Outpatient clinic visit (Day 14)
* Week 4: Telephone visit (Day 21)
* Week 5: 24 to 48-hour in-clinic stay (Day 28)
* Week 6: Follow-up visit (Day 35) Disclosure Statement: The study consists of two cohorts, each with a parallel-group design and two arms, with participants blinded to treatment allocation.

Number of Participants:

The study will randomise approximately 36 participants in total. Cohort A: Approximately 75 participants with presumed MASH/NASH with fibrosis will be screened such that approximately 18 participants will be randomised. Twelve participants will be randomised to receive AZD2389 and 6 participants will receive placebo. Cohort B: Approximately 75 participants with SLD with advanced fibrosis including compensated cirrhosis will be screened such that approximately 18 participants will be randomised. Twelve participants will be randomised to receive AZD2389 and 6 participants will receive placebo

ELIGIBILITY:
Key inclusions:

* Males/females aged ≥ 18 years
* Indications: Presumed MASH (cohort A) or other steatotic liver disease (cohort B) with fibrosis
* No significant change in weight over the last 6 months
* Barrier contraceptives use by males
* Capable of informed consent
* Judged to be suitable for study by investigator

Key exclusions:

* A condition that could put the participant at risk, influence the participant's ability to participate in the trial, interfere with evaluation of the study intervention or affect the interpretation of the results
* Other causes of liver disease which are not the principal inclusion criteria for each cohort
* Significant elevations in liver blood tests or platelets <140 x10^9/L
* Decompensated liver disease, hepatobiliary cancer or listing for liver transplantation
* Bleeding disorders or major bleeding risk
* HIV infection or hepatitis B infection
* Clinically significant cardiovascular (e.g. severe ischaemic heart disease, severe heart failure or cardiac dysrhythmia) or cerebrovascular disease within the past 3 months
* Stage 2 hypertension
* eGFR <60ml/min/1.73m2
* Clinically significant gastrointestinal disease which can affect the interpretation of pharmacokinetic, safety, and tolerability data
* Skin disorders or ongoing wound healing
* Psychiatric disorders which may negatively affect participation in the trial.
* Females of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Reported quantity and severity of adverse events (AEs) following oral administration of AZD2389 | Up to and including day 35 (from pre-screening to follow-up visit)
  Reporting frequency and severity of AEs based on qualifying symptoms, signs, abnormalities in measured values, or other diagnoses as identified by investigator
Number of participants with observed changes in blood pressure against baseline mmHg value | Up to and including Day 35 (from pre-screening to follow-up visit)
  Assess blood pressure level (with systolic and diastolic pressure) in mmHg
Number of participants with observed changes in heart rate (BPM) against baseline value | Up to and including day 35 (from pre-screening to follow-up visit)
  Pulse rate measured in beats per minute (BPM)
Number of participants with observed changes in Sp02 oxygen values against baseline measurement | Up to and including day 35 (from pre-screening to follow-up visit)
  Sp02 oxygen saturations measured by percentage
Number of participants with observed changes in body temperature against baseline value | Up to and including day 35 (from pre-screening to follow-up visit)
  Body temperature measured in degrees Celsius
Number of participants with observed changes in respiratory rate against baseline value | Up to and including day 35 (from pre-screening to follow-up visit)
  Respiratory rate measured in respirations per minute
Number of participants with identified abnormalities in results of 12-lead safety electrocardiograms (ECG) | Up to and including day 35 (from pre-screening to follow-up visit)
  12-lead safety ECG (PR interval, QRS complex, ST interval, T wave)
Number of participants with changes in physical baseline values identified during physical examinations | Up to and including day 35 (from pre-screening to follow-up visit)
  Physical examinations will include assessment of general appearance, skin, head and neck (including ears, eyes, nose and throat), lymph nodes, thyroid, musculoskeletal (including spine and extremities) and neurological symptoms (examination of the participants' feet to observe skin integrity, circulation, and presence of any neuropathy).
Number of participants with abnormal laboratory test results detected in blood samples | Up to and including day 35 (from pre-screening to follow-up visit)
  Hematology - Platelets (x10^9/L) Clinical Chemistry - ALT (U/L), AST (U/L), ALP (U/L) Coagulation - INR Fibrinolysis - D-dimer (ng/mL fibrinogen-equivalent units)
Number of participants with abnormal laboratory results detected in urine samples | Up to and including day 35 (from pre-screening to follow-up visit)
  Urinalysis - Paper chromatography
Number of participants with visible changes (against baseline observations) to the condition of abdominal organs as identified by FibroScan imaging | Up to and including Day 35 (from pre-screening to follow-up visit)
  FibroScan (VCTE) ultrasound imaging will measure a participant's level of LSM (liver stiffness), CAP (amount of fat in the liver), and/or SSM (spleen stiffness).

SECONDARY OUTCOMES:
To evaluate the effect of AZD2389 on plasma FAP activity following oral administration of AZD2389 in participants with CLD and hepatic fibrosis | From Day 1 to Day 35
  Inhibition of FAP activity at Days 1, 7, 14, 28, and follow-up (calculated as change and percentage change in FAP activity against baseline) compared to placebo
Maximum Plasma Concentration (Cmax) detected in blood sample | From Day 1 to Day 35
  Maximum Plasma Concentration (Cmax)
Time to Maximum Concentration (Tmax) as detected in blood sample | From Day 1 to Day 35
  Time to Maximum Concentration (Tmax)
Area Under the Concentration-time Curve to the Last Measurable Concentration (AUClasta) as detected in blood sample | From Day 1 to Day 35
  Area Under the Concentration-time Curve to the Last Measurable Concentration (AUClasta)
Area Under the Concentration-time Curve Extrapolated to Infinity (AUCinf) as detected in blood sample | From Day 1 to Day 35
  Area Under the Concentration-time Curve Extrapolated to Infinity (AUCinf)
Area Under the Concentration-time Curve Over a Dosing Interval (AUCtau) as detected in blood sample | From Day 1 to Day 35
  Area Under the Concentration-time Curve Over a Dosing Interval (AUCtau)
Terminal Half-life (t1/2λz) as detected in blood sample | From Day 1 to Day 35
  Terminal Half-life (t1/2λz)
Apparent Volume of Distribution (Vz/F) as detected in blood sample | From Day 1 to Day 35
  Apparent Volume of Distribution (Vz/F)
Apparent Clearance (CL/F) as detected in blood sample | From Day 1 to Day 35
  Apparent Clearance (CL/F)
Temporal Change Parameter (TCP) as detected in blood sample | From Day 1 to Day 35
  Temporal Change Parameter (TCP)
Cmax Accumulation Ratio (Rac Cmax) as detected in blood sample | From Day 1 to Day 35
  Cmax Accumulation Ratio (Rac Cmax)
AUC Accumulation Ratio (Rac AUC) as detected in blood sample | From Day 1 to Day 35
  AUC Accumulation Ratio (Rac AUC)
Renal Clearance (CLR) as detected in blood sample | From Day 1 to Day 35
  Renal Clearance (CLR)
Amount of Drug Excreted in Urine (Ae) as detected in urine sample | From Day 1 to Day 35
  Amount of Drug Excreted in Urine (Ae)
Fraction of Drug Excreted in Urine (Fe) as detected in urine sample | From Day 1 to Day 35
  Fraction of Drug Excreted in Urine (Fe)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Research Site, Chandler, Arizona
  - Research Site, Rialto, California
  - Research Site, Atlanta, Georgia
  - Research Site, Morehead City, North Carolina
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
- Research Site, San Juan, Puerto Rico
- Research Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/